CLINICAL TRIAL: NCT03536130
Title: Multicenter Randomized Study on Comparison Between Electronic and Traditional Chest Drainage Systems
Brief Title: Comparison Between Electronic and Traditional Chest Drainage Systems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Padova (Other)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Vito Fazzi Hospital (Unknown); Monaldi Hospital (Other)
Responsible Party: Principal Investigator, PROF. GIUSEPPE MARULLI, MD, PhD, University Hospital Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4013/AO/16
Record Dates: First submitted 2018-04-20; First posted 2018-05-24 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Lung Cancer
Keywords: chest tube, lung resection, air leakage
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Allocation: randomization 1 to 1 Endpoint classification: efficacy study Masking: Open label Intervention model: parallel assignment Primary purpose: supportive care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic chest drainage system (Experimental): Patients in the intervention arm are connected to Drentech Palm Evo with single standard chest tube (28 Ch) immediately after closure of the chest. Patients with digital devices are managed by setting the pump to -20 cmH2O until the morning of postoperative day (POD) 1 and then setting the pump on physiologic mode (0 cmH2O) thereafter.
  Interventions: Device: Electronic chest drainage system
- Traditional device (No Intervention): Patients in the no intervention (traditional) arm are connected to traditional drain system with single standard chest tube (28 Ch) immediately after closure of the chest. Patients with traditional devices (requiring connection to wall suction) are managed by applying suction (-20 cmH2O) until the morning of POD 1 and are subsequently disconnected from suction thereafter.

INTERVENTIONS:
Device: Electronic chest drainage system — Patients in the intervention arm are connected to Drentech Palm Evo with single standard chest tube (28 Ch) immediately after closure of the chest. Patients with digital devices are managed by setting the pump to -20 cmH2O until the morning of postoperative day (POD) 1 and then setting the pump on physiologic mode (0 cmH2O) thereafter. Management of chest tube drainage and decision for chest tube removal will be dictated by clinical signs, symptoms and surgeon preference following standard clinical practice of general thoracic patients
  Arms: Electronic chest drainage system

SUMMARY:
This study is designed to compare the electronic chest drainage system (Drentech Palm Evo) with the traditional system, both already in use in the clinical practice, in a cohort of patients who received thoracoscopic lobectomy. This study is not evaluating safety or efficacy of these systems.

This study's primary aim is to determine if the use of a digital chest system compared with a traditional system reduce the duration of chest drainage and length of hospital stay. Moreover, the investigators aim to quantify the variability of results regarding the subjective observer evaluation of active air leaks (through the traditional system) compared with the objective data registered by the digital system.

Finally the investigators want to evaluate whether it is possible through the digital device to distinguish an active air leak from a pleural space effect by the evaluation of intrapleural differential pressure and to identify potential predictors of prolonged air leaks.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to read, understand and provide written informed consent
* Patients undergoing thoracoscopic lobectomy
* Age 18 - 80 years
* Gender: both
* Estimated life expectancy of at least 6 months.
* Tumour considered potentially resectable by R0 surgery
* Adequate respiratory function for surgery.
* Must have signed and dated an informed consent form (ICF), before performance of any study-specific procedures or tests. Subjects must be fully informed about their illness and the investigational nature of the study protocol.

Exclusion Criteria:

* Patients requiring ICU care with mechanical ventilation
* Patients needing reintervention during postoperative care
* Patients requiring a thoracotomy
* Tumour considered potentially resectable by incomplete surgical resection with microscopic residual disease (R1) or gross residual disease (R2).
* Evidence of extra-thoracic disease.
* Major thoracic surgical procedure before enrolment.
* Any other significant co-morbid condition that, in opinion of the investigator, would impair study participation or cooperation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Estimated)
Dates: Start 2017-04-04 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Duration of chest drainage | from date of surgery to date of chest tube removal, assessed up to 8 days
Post-operative hospital length of stay | from date of surgery to date of hospital discharge, assessed up to 8 days
Evaluation of the degree of concordance between the subjective observer evaluation of active air leaks compared with the objective data registered by the digital system in the patients with electronic chest drainage system | from date of surgery to date of chest tube removal, assessed up to 8 days

SECONDARY OUTCOMES:
Evaluation of intrapleural differential pressure in case of active air leak and in case of pleural space effect | from date of surgery to date of chest tube removal, assessed up to 8 days
Identification of potential predictors of prolonged air leaks through the analysis of the data registered by the digital system | from date of surgery to date of chest tube removal, assessed up to 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Marulli, MD, PhD, Principal Investigator — Thoracic Surgery Unit - University Hospital of Padova
Locations (4):
- Italy (4):
  - Thoracic Surgery Unit, Vito Fazzi Hospital, Lecce
  - Thoracic Surgery Unit, Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, University of Milan, Italy, Milan
  - Thoracic Surgery Unit, Monaldi Hospital, Napoli
  - Thoracic Surgery Unit - University of Padova, Padua

REFERENCES:
- [Derived] Mendogni P, Tosi D, Marulli G, Comacchio GM, Pieropan S, Rossi V, Brascia D, Andriolo LG, Imbriglio G, Bonitta G, Lopez C, Rea F, Nosotti M. Multicenter randomized controlled trial comparing digital and traditional chest drain in a VATS pulmonary lobectomy cohort: interim analysis. J Cardiothorac Surg. 2021 Jul 5;16(1):188. doi: 10.1186/s13019-021-01567-y. PMID 34225743
- [Derived] Marulli G, Comacchio GM, Nosotti M, Rosso L, Mendogni P, Natale G, Andriolo L, Imbriglio G, Larocca V, Brascia D, Rea F. Multicenter randomized study on the comparison between electronic and traditional chest drainage systems. Trials. 2019 Dec 16;20(1):730. doi: 10.1186/s13063-019-3811-8. PMID 31842974